CLINICAL TRIAL: NCT01623232
Title: MAS-1 Adjuvanted Compared to Unadjuvanted Influenza Vaccines in the Elderly
Acronym: CCTA #0005
Status: Withdrawn | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: FDA hold on the project
Sponsor: US Department of Veterans Affairs (U.S. Federal Agency)
Collaborators: St. Louis University (Other)
Responsible Party: Sponsor
Organization: VA Office of Research and Development (U.S. Federal Agency)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: CLIN-07-11S; 1 I01 CX000633-01 (Other Grant/Funding Number: VA)
Record Dates: First submitted 2012-06-15; First posted 2012-06-19 (Estimated); Last update posted 2012-09-26 (Estimated); Status verified 2012-09

CONDITIONS: Influenza Vaccines; Aged
Keywords: vaccine; influenzavirus A; influenzavirus B; adjuvant
MeSH Terms: conditions — Influenza, Human

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- adjuvant plus 1 �g of HA antigen (Experimental): MAS-1-adjuvant-formulated influenza vaccine, at three HA antigen dose levels containing 1 �g of HA antigen
  Interventions: Biological: MAS-1 adjuvant and influenza HA antigen
- adjuvant plus 3 �g of HA antigen (Experimental): MAS-1-adjuvant-formulated influenza vaccine, at three HA antigen dose levels containing 3 �g of HA antigen
  Interventions: Biological: MAS-1 adjuvant and influenza HA antigen
- adjuvant plus 5 �g of HA antigen (Experimental): MAS-1-adjuvant-formulated influenza vaccine, at three HA antigen dose levels containing 5 �g of HA antigen
  Interventions: Biological: MAS-1 adjuvant and influenza HA antigen
- licensed influenza vaccine (Active Comparator): licensed, inactivated, standard dose influenza vaccine without adjuvant
  Interventions: Biological: standard dose, inactivated trivalent influenza vaccine (TIV)

INTERVENTIONS:
Biological: MAS-1 adjuvant and influenza HA antigen — Vaccines will be administered IM in the deltoid muscle. HA antigen of each of three viral strains at doses of 1 micrograms, 3 micrograms, or 5 micrograms per viral strain adjuvanted with MAS-1 adjuvant and as nonadjuvanted standard dose TIV will be tested.
  1. Treatment Group 1:each 0.3 mL dose will be administered as an emulsion containing 0.186 grams of MAS-1 oil vehicle and 1 micrograms HA of each of three viral strains in 0.08 mL sterile phosphate buffered saline (PBS).
  2. Treatment Group 2:each 0.3 mL dose will be administered as an emulsion containing 0.186 grams of MAS-1 oil vehicle and 3 micrograms HA of each of three viral strains in 0.08 mL sterile PBS.
  3. Treatment Group 3:each 0.3 mL dose will be administered as an emulsion containing 0.186 grams of MAS-1 oil vehicle and 5 micrograms HA of each of three viral strains in 0.08 mL sterile PBS.
  Other Names: MER4101
  Arms: adjuvant plus 1 �g of HA antigen; adjuvant plus 3 �g of HA antigen; adjuvant plus 5 �g of HA antigen
Biological: standard dose, inactivated trivalent influenza vaccine (TIV) — Vaccine will be administered IM in the deltoid muscle. HA antigen of each of three viral strains as nonadjuvanted standard dose TIV will be tested.
  4. Treatment Group 4:0.5 mL dose of licensed, unadjuvanted, standard dose influenza virus vaccine with 15 micrograms HA of each of 3 viral strains.
  Arms: licensed influenza vaccine

SUMMARY:
This is a Phase 1,2 randomized, double-blind, multi-center, clinical trial, in participants aged 65 years and older, evaluating the immunogenicity and safety of a water-in-oil emulsion adjuvant (MAS-1 adjuvant, Mercia Pharma, Inc, Scarsdale, NY) combined with each of the three reduced HA antigen dose levels of trivalent influenza virus vaccine compared with licensed, unadjuvanted, standard dose trivalent virus (TIV). Immunogenicity for each of the three viral strains (A/H1N1, A/H3N2, and B virus) in the concurrent influenza seasonal vaccine will be assessed.

DETAILED DESCRIPTION:
Many VA patients are at-risk for complications from influenza because of advanced age and underlying chronic diseases. A more effective influenza virus vaccine is needed in older patient populations and high antibody levels are correlated with protection. Vaccine dose-sparing to maximize the number of doses available is a public health goal. The combination of influenza vaccine antigens with an adjuvant could help improve the vaccine. This study will be a phase 1, 2 randomized, observer-blind, multi-center, clinical trial, in patients aged 65 years and older, evaluating the immunogenicity and safety of a water-in-oil emulsion adjuvant (MAS-1) combined with each of three reduced influenza hemagglutinin (HA) antigen dose levels of trivalent influenza virus vaccine compared to unadjuvanted, standard dose trivalent influenza virus vaccine (TIV). Immunogenicity for each of the three viral strains (A/H1N1, A/H3N2, and B virus) in the concurrent seasonal influenza vaccine will be assessed. The hypothesis is that adjuvanted influenza virus vaccine (using reduced doses of influenza HA antigen containing 1 g, 3 g and 5 g of HA) has superior immunogenicity compared to unadjuvanted, standard dose trivalent influenza virus vaccine (containing 15 g HA antigen) for each of three viral strains, and the adjuvanted vaccine has an acceptable safety profile. The primary objectives are to demonstrate 1) acceptable safety for influenza virus vaccine, adjuvanted with MAS-1 compared to unadjuvanted, standard dose TIV, and 2) improved immunogenicity of the adjuvanted influenza virus vaccine compared to unadjuvanted, standard dose TIV for each of the three viral strains. Immunogenicity will be measured by hemagglutination inhibition (HAI) antibody titers. The primary measure of immunogenicity is the seroconversion rate at 1 month post-vaccination for each viral strain. Secondary and exploratory immunogenicity objectives include the seroprotection rate (defined as the proportion of subjects with a post-vaccination HAI antibody titer > 1:40 for a viral strain) at 1, 3 and 6 months post-vaccination for each viral strain; the geometric mean titers (GMTs) of HAI antibody and ratio of GMTs pre-vaccination and at 1, 3 and 6 months post-vaccination between the four vaccine groups for each viral strain; and the geometric mean fold increase (GMFI) at 1, 3 and 6 months post-vaccination compared to pre-vaccination (i.e., GMT of the post-vaccination values divided by the GMT of the pre-vaccination value) for each virus strain within each of the four vaccine groups. The study population of 160 subjects (40 per vaccine group) who provide informed consent and meet eligibility criteria will be enrolled at four clinical sites. Subjects who meet the entry criteria for the study will be randomly assigned to receive one of the three adjuvanted influenza virus vaccine dose levels or unadjuvanted, standard dose TIV. Randomization will be stratified by clinical site (4 sites) and age (65-74 years old or 75 years old). Vaccine preparation will be performed at point-of-use by the site pharmacists according to a standardized procedure. Administration of vaccine will be performed by an unblinded vaccine administrator. Study assessments will be performed by blinded study personnel. Subjects will also be blinded to treatment assignment. Study subjects will each participate for a total of 12 months post-vaccination. The whole study duration of 32 - 32.5 months is expected to include 6 months of startup, 8 - 10 weeks of enrollment, 12 months of follow-up post-vaccination and 12 months of study closure and data analysis. If the objectives of this study are achieved and the hypothesis is correct, the adjuvanted influenza virus vaccine at one or more of the reduced HA antigen doses will induce an improved HAI antibody response compared to unadjuvanted, standard dose TIV with an acceptable safety profile. Results of this trial will inform the design of future clinical trials studying adjuvanted influenza virus vaccines utilizing this novel water-in-oil adjuvant emulsion that could include dose-finding studies for the optimal amount of adjuvant combined with one HA antigen dose, and larger phase 2 and 3 clinical trials.

ELIGIBILITY:
Inclusion Criteria:

Participants must meet all of the following inclusion criteria at Screening/Baseline to participate in this study:

1. Ambulatory persons aged at least 65 years or older on the day of enrollment. Participants will be considered ambulatory if they are not institutionalized, bedridden, or homebound.
2. Written informed consent form and Authorization to Obtain and Release Protected Health Information (HIPAA) form signed.
3. Medically stable. Participants may have clinically stable underlying chronic conditions such as, but not limited to hypertension, diabetes, congestive heart failure, ischemic heart disease, or chronic lung disease, but their symptoms/signs must be controlled, as judged by the investigator, based on physical examination and medical history. Participants with pre-existing stable disease, defined as disease not requiring significant change in therapy or hospitalization for worsening disease 4 weeks before receipt of the test article, are eligible.
4. Body Mass Index (BMI)<40
5. Normal ranges for safety labs including:

   * WBC count 3,600 - 11,200 cells/mm3
   * Platelets: 150,000-450,000/mm3
   * Hemoglobin >sex-specific institutional lower limit of normal (Female 11 g/dL and Male 12.5 g/dL).
   * Chemistry Panel: ALT, AST, total bilirubin <1.1 times and CPK <1.25 times the upper limit of normal for the study; glucose 65 to 100 mg/dL; creatinine 0.40 to 1.40 mg/dL
   * Absolute neutrophil, lymphocyte and eosinophil counts are within the study normal range.
   * Normal urine dipstick: negative or trace urine protein, negative or trace urine blood.
6. Able to attend all scheduled visits and to comply with all trial procedures.

Exclusion Criteria:

Participants who meet any of the exclusion criteria at Screening/Baseline will be excluded from study participation. Participants will not be able to participate if they have:

1. Systemic hypersensitivity to eggs, chicken proteins, or any of the other vaccine components, or a history of a life-threatening reaction to TIV or a vaccine containing any of the same substances.
2. History of congenital or acquired immunodeficiency, Human Immunodeficiency Virus infection, hepatitis C or B virus infection, or autoimmune disease, or immunosuppressive therapy or radiation therapy in the preceding six months.
3. Systemic corticosteroid therapy, as follows:

   * Continuous use with a dosage equivalent to >15 mg per day of oral prednisone for 90 days preceding vaccination.
   * Sporadic use with a dosage equivalent to >40 mg per day of oral prednisone for >14 consecutive days in the 90 days preceding vaccination.
4. Neoplastic disease or any hematologic malignancy (except localized skin or prostate cancer that is stable at the time of vaccination in the absence of therapy, and history of neoplastic disease but disease-free for 5 years).
5. Current alcohol abuse or drug addiction that may interfere with trial procedures.
6. Receipt of blood or blood-derived products in the past three months.
7. Receipt of influenza vaccine in the past six months.
8. Receipt of any other vaccine in the past four weeks.
9. Planned receipt of another vaccine in the four weeks following the trial vaccination.
10. Planned participation in another clinical trial during the present trial period. Concomitant participation in an observational trial (not involving drugs, vaccines, or medical devices) is acceptable.
11. Thrombocytopenia or bleeding disorder contraindicating IM vaccination. Anticoagulation is only a relative contraindication to IM vaccine injections (39). Exclusion from participation on this basis is at the discretion of the participant and the investigator after full discussion of the risks.
12. History of Guillain-Barr syndrome.
13. An acute febrile illness within 24 hours prior to vaccination. Vaccination will be deferred until the participant has been afebrile for at least 24 hours.
14. Signs and symptoms of an acute infectious respiratory ill

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 0 (Actual)
Dates: Start 2012-10; Primary Completion 2013-11 (Estimated); Study Completion 2014-06 (Estimated)

PRIMARY OUTCOMES:
safety | 12 months
  Participants with at least one vaccine-related adverse event (AE) from the following four categories: solicited AEs, unsolicited AEs, serious AEs, and abnormal safety labs for severity grade 2 or higher, grade 3 only, and grade 4 or 5.

SECONDARY OUTCOMES:
immunogenicity | 6 months
  The primary immunogenicity outcome is the seroconversion rate at 1 month (day 28) post-vaccination for each of the three virus strains in each vaccine group. Seroconversion rate at 1 month is defined as the proportion of participants with either a pre-vaccination HAI antibody titer <1:10 and a post-vaccination antibody titer = 1:40, or a pre-vaccination HAI antibody titer = 1:10 and a minimum four-fold rise in post-vaccination antibody titer.
immunogenicity | 1 month
  The seroprotection rate at 1 month (day 28) post-vaccination for each of the three virus strains in each vaccine group. Seroprotection is defined as the proportion of participants with post-vaccination antibody titer of 1:40 or greater.
immunogenicity | 1 month
  The geometric mean titers of antibody and ratios of geometric mean antibody titers at 1 month (28 days) post-vaccination for each virus strain and vaccine group.
immunogenicity | 6 months
  The seroprotection rates up to 6 months post-vaccination for each virus strain and vaccine group.
immunogenicity | 6 months
  The rates of antibody titers at serum dilutions of at least 1:80, at least 1:160, and at least 1:320.
immunogenicity | 6 months
  The geometric mean antibody titers and ratios of geometric mean antibody titers up to 6 months post-vaccination for each virus strain and vaccine group.
safety | 12 months
  Participants in each vaccine group experiencing an individual adverse event (AE) by severity grade, relatedness to vaccine, for solicited AEs, unsolicited AEs, serious AEs and abnormal safety labs.
safety | 12 months
  Participants in each vaccine group experiencing at least one abnormal symptom with any severity grade, grade 2 or higher, grade 3 or higher, and grades 4 and 5, by relatedness to vaccine, for solicited adverse events (AE), serious AEs and safety labs.

CONTACTS AND LOCATIONS:
Overall Officials: Geoffrey J. Gorse, MD, Principal Investigator — St. Louis VA Medical Center John Cochran Division, St. Louis, MO
Locations (4):
- United States (4):
  - VA Palo Alto Health Care System, Palo Alto, CA, Palo Alto, California
  - Iowa City VA Health Care System, Iowa City, IA, Iowa City, Iowa
  - Minneapolis VA Health Care System, Minneapolis, MN, Minneapolis, Minnesota
  - St. Louis VA Medical Center John Cochran Division, St. Louis, MO, St Louis, Missouri